CLINICAL TRIAL: NCT04657718
Title: CLAIM: Using the KODEX-EPDTM System to Guide PaCing Lead Placements, A First In Man Study
Brief Title: CLAIM: Using the KODEX-EPD System to Guide PaCing Lead Placements, A First In Man Study.
Acronym: CLAIM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study never started - clinical strategy changed
Sponsor: EPD Solutions, A Philips Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIPS635841
Record Dates: First submitted 2020-11-17; First posted 2020-12-08 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2020-06

CONDITIONS: Cardiac Arrhythmia
Keywords: Pacing Lead implantation; KODEX-EPD; CRT; His bundle pacing; LBBP
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All subjects (Other): The KODEX-EPD system will be used in combination with leads to image during all procedures.
  Interventions: Device: KODEX-EPD system

INTERVENTIONS:
Device: KODEX-EPD system — Cardiac pacing leads implantation for PM, ICD, CRT, HBP and LBBP

SUMMARY:
Prospective, multi-center (2-3 sites), non-randomized, open label, single arm 3 phase study:

1. Phase 1 or Evaluation Phase: Where the KODEX-EPD System will be used to exclusively monitor the entire implantation procedure; the KODEX-EPD system will not be used for guidance during the lead implantation workflow.
2. Phase 2 - KODEX-EPD-assisted Phase: Where the KODEX-EPD system will be used for cardiac imaging acquisition, guidance during lead implantation in conjunction with fluoroscopic imaging
3. Phase 3 - KODEX-EPD-guided Phase: Where the KODEX_EPD System will be used as the leading imaging modality during the lead implantation workflow. Fluoro can be used;

   * up until the part of the lead implantation workflow that is the scope of this investigation.
   * As a bailout, when the operator declares failure to attempt.

ELIGIBILITY:
Patients scheduled to undergo lead placement for cardiac pacing. Subjects who meet all eligibility criteria and give written informed consent will be enrolled in the study.

Inclusion Criteria:

1. Subject must be aged >18 years.
2. Subject must have signed a written iInformed Cconsent form to participate in the study, prior to any study related procedures.
3. Subject must be willing to comply with the protocol requirements.
4. Subject is scheduled for a de novo pacing lead implantation or system upgrade .

Exclusion Criteria:

1. Patients for whom previous CRT or conduction pacing implantation has failed.
2. Patients considered for leadless cardiac pacing system.
3. Patients undergoing a system revision for infection or malfunction.
4. Patients undergoing planned, urgent or emergency lead revision or lead extraction.
5. Subjects who have received or will receive an experimental drug or used an experimental medical device within 30 days before the planned start of treatment.
6. Patients included in a clinical registry or clinical trial for an investigational product.
7. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Incidence of intra -and Perioperative complications | 3 months
  Incidence rate of intra -and Perioperative complications (bleeding, hematoma, cardiac tamponade, cardiac perforation , appearance of hemodynamic relevant arrhythmias requiring intervention)
Primary Feasibility Endpoint - Ability of imaging with permanent implantable leads and guidewires. | time of procedure - 2-5 hours
  The successful use of permanent implantable leads and guidewires for imaging with KODEX - EPD. Assessment of the ability of the KODEX-EPD system to create real time 3D images of the anatomy of the heart.

SECONDARY OUTCOMES:
Right heart image | time of procedure - 2-5 hours
  Number of patients in whom it is possible to construct a right heart endocardial image, including visualization of right atrial appendage, tricuspidal valve, coronary sinus ostium, and coronary veins in case of CRT device implantation.
Lead implantation adjusted with Fluoroscopy | time of procedure - 2-5 hours
  Number of patients in whom lead implantation needs to be fluoroscopically adjusted after KODEX-EPD-guided implantation because of 1) inability to overcome anatomical obstacles; 2) mechanical instability including spontaneous dislodgement; 3) unsatisfactorily electrical parameters.
Fluoroscopy time | time of procedure - 2-5 hours
  Total fluoroscopy time
Use of Contrast | time of procedure - 2-5 hours
  Total amount of contrast used, if any.
Procedure Time - per lead | time of procedure - 2-5 hours
  Time to final placement, for each implanted lead (from lead introduction into sheath to final placement)
Procedure Time - all leads | time of procedure - 2-5 hours
  Total lead(s) implantation time
Total procedure time | time of procedure - 2-5 hours
  Total implantation time (skin-to-skin)
Fluoroscopy dose | time of procedure - 2-5 hours
  Total fluoroscopy dose

IPD SHARING:
Plan to Share IPD: No